CLINICAL TRIAL: NCT06008548
Title: A New Conception About Individualized Treatment Allocation for HCC-Using Machine Learning
Brief Title: A New Conception About Individualized Treatment Allocation for HCC
Acronym: PTA4HCC
Status: Completed | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Collaborators: Air Force Military Medical University, China (Other); Army Medical University, China (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Sun Yat-sen University (Other); Shaanxi Provincial People's Hospital (Other); Xijing Hospital (Other); Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: liulei
Record Dates: First submitted 2023-04-02; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: HCC; Transarterial Chemoembolization; Resection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TACE group: Incorporated HCC patients underwent TACE therapy.
  Interventions: Procedure: TACE
- Liver resection group: Incorporated HCC patients underwent liver resection therapy.

INTERVENTIONS:
Procedure: TACE
  Groups: TACE group

SUMMARY:
The current guidelines on hepatocellular carcinoma (HCC) aimed to build effective prognostic stratification strategies to guide therapeutic allocation; however, the current guidelines did not consider the simultaneous comparison of distinct therapies in similar populations. Here, the investigators aimed to develop and validate a new, integrated prognostic scheme for HCC patients using artificial intelligence (AI) to simulate the survival outcomes of patients allocated to different treatments.

DETAILED DESCRIPTION:
Given that liver resection (LR) and transarterial chemoembolization (TACE) are the mainstay curative and palliative therapies for HCC, respectively, patients who underwent LR or TACE were included in the study. Various prognostic AI algorithms were modeled using data from a large multi-institutional cohort, where LR and TACE were considered independent factors. The C-index, Brier score (BS), and area under the receiver operating characteristic curve (auROC) were calculated to estimate the AI models.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with HCC
* Receiving LR or TACE therapy
* Complete clinical information
* Preserved liver function (Child-Pugh Score [CPS] ≤ 7)
* PS 0-1

Exclusion Criteria

* Vascular invasion or extrahepatic spread;
* Ecompensated liver cirrhosis ;
* Younger than 18 years;
* Duration of follow-up of fewer than 30 days.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January 2010 and October 2021, a total of 4991 consecutive HCC patients receiving LR or TACE from 15 Chinese tertiary hospitals were retrospectively screened. HCC was diagnosed based on either imaging or pathological results as previously described
Sampling Method: Probability Sample
Enrollment: 4991 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 years
  Overall survival (OS) was defined as the time interval between initial TACE or LR and all-cause death. Patients who survived up to the last follow-up date

CONTACTS AND LOCATIONS:
Overall Officials: Lei Liu, doctor, Study Director — Tangdu Hospital-Air Force Medical University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT06008548/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT06008548/ICF_001.pdf